CLINICAL TRIAL: NCT02156570
Title: An Interferon Sparing Strategy of Sofosbuvir Plus Ribavirin for the Treatment of Recently Acquired Hepatitis C Infection
Brief Title: DAA-based Therapy for Recently Acquired Hepatitis C II (DAA = Directly Acting Antiviral)
Acronym: DARE-C II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHCRP1206
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Acute/early chronic; Recently acquired; Directly acting antiviral therapy; Sofosbuvir; Ribavirin
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome | interventions — Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sofosbuvir and ribavirin (Experimental): Sofosbuvir tablet 400 mg daily Ribavirin tablet weight based dosing (1000mg <75 kg, 1200mg >/= 75kg) daily
  Treatment will be for 6 weeks in all participants.
  Interventions: Drug: Sofosbuvir and ribavirin

INTERVENTIONS:
Drug: Sofosbuvir and ribavirin — Sofosbuvir 400mg daily plus weight-based dosing ribavirin (1000mg <75kg, 1200mg >/= 75 kg) Treatment will be for 6 weeks in all participants.
  Other Names: Sovaldi; Copegus

SUMMARY:
The purpose of the study is to examine whether patients who have acute or early chronic hepatitis C virus (HCV) infection can be treated effectively and safely with an interferon-sparing regimen that combines a new direct acting antiviral drug (sofosbuvir) with one of the standard treatments for chronic hepatitis C (ribavirin). In particular, this study will investigate whether treatment of acute or early chronic HCV can be shortened. The study will assess efficacy by looking at the proportion of people who clear the virus (have no virus detectable in their blood) at the end of treatment, and 1, 3 and 6 months after treatment.

The hypothesis is that short course (6 weeks) dual therapy using sofosbuvir and RBV will result in successful virological eradication in the majority (≥80%) of subjects treated for recently acquired HCV.

DETAILED DESCRIPTION:
To evaluate the efficacy, safety and acceptability of an interferon-sparing strategy with sofosbuvir and ribavirin for the treatment of recently acquired HCV infection.

An open label single arm multicentre study Treatment of participants: Sofosbuvir 400mg daily with weight based ribavirin (1000mg <75 kg, 1200mg >/= 75kg) Duration of treatment will be 6 weeks for all subjects followed by 52 weeks of observational follow-up Total study duration = 58 weeks Primary endpoint: SVR 12

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Male and female patients aged 18 years and above
* Willing to use two effective methods of contraception during the treatment period and 24 weeks post.
* HBsAg negative
* Detectable HCV RNA at screening (>10,000 IU/ml), and in the opinion of the investigator is unlikely to demonstrate spontaneous viral clearance
* Compensated liver disease (Child-Pugh A)
* Negative pregnancy test at screening and 24 hours prior to first dose of study drugs
* Medically stable on the basis of physical examination, medical history and vital signs
* Adequate English to provide reliable responses to the study questionnaires
* Recent hepatitis C infection, as defined by: A) i) First anti-HCV Ab or HCV RNA positive within the previous 6 months and ii) Documented anti-HCV Ab negative within the 24 months prior to anti-HCV antibody positive result, OR B) i) First anti-HCV Ab or HCV RNA positive within the previous 6 months and ii) acute clinical hepatitis (jaundice or ALT> 10 X ULN) within the previous 12 months prior to first positive HCV antibody or HCV RNA, with no other cause of acute hepatitis identifiable

If co-infection with HIV is documented, the subject must meet the following criteria:

* Antiretroviral (ARV) untreated for >8 weeks preceding screening visit with CD4 T cell count >500 cells/mm3 OR
* On a stable ARV regimen for >8 weeks prior to screening visit, with CD4 T cell count >200 cells/mm3 and an undetectable plasma HIV RNA level.

Exclusion Criteria:

* Standard exclusions to RBV therapy
* Pregnancy/lactation or male subjects whose female partners are pregnant
* Subject has a history of decompensated liver disease: history of ascites, hepatic encephalopathy, or bleeding oesophageal varices, and/or any of the following screening laboratory results: a.INR of ≥1.5; Serum albumin <3.3 g/dL; Serum total bilirubin >1.8 times upper limit of normal, unless isolated in subjects with Gilbert's syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
SVR 12 | 12 weeks post treatment
  Proportion of patients with undetectable HCV RNA by TaqMan 12 weeks after therapy completion (SVR 12 - Week 18)

SECONDARY OUTCOMES:
SVR 24 | 24 weeks post treatment
  Proportion of patients with undetectable HCV RNA by TaqMan 24 weeks after therapy completion (SVR 24 - Week 30)

OTHER OUTCOMES:
End of treatment response | End of treatment week 6
  Proportion of patients with undetectable HCV RNA at end of therapy (ETR - week 6)
SVR 4 | 4 weeks post treatment
  Proportion of patients with undetectable HCV RNA by TaqMan 4 weeks after therapy completion (SVR 4 - Week 10)
Follow up 1 year | 1 year post treatment
  Proportion of patients with undetectable HCV RNA at end of study follow-up (FU1 - Week 58)
Undetectable HCV RNA | Week 1, 2, 3 and 4 of treatment
  Proportion of patients with undetectable HCV RNA at weeks 1, 2, 3 and 4
Indicators of toxicity (ALT, HB, Neutrophils, Platelets) | Baseline until week 4 of treatment
  To evaluate indicators of toxicity (ALT, HB, Neutrophils, Platelets) during therapy
Plasma ribavirin levels and haemoglobin | Baseline to week 4 of treatment
  To correlate plasma ribavirin levels with treatment outcome and changes in haemoglobin during therapy
Incidence of reinfection | End of treatment until follow up 1 year
  Incidence of reinfection after documented SVR

CONTACTS AND LOCATIONS:
Overall Officials: Gail Matthews, MbChB FRACP, Principal Investigator — Kirby Institute
Locations (5):
- Australia (4):
  - St Vincent's Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
- Auckland City Hospital, Auckland, Grafton, New Zealand

REFERENCES:
- See also: UNSW Kirby Institute for infection and immunity in society Homepage — http://www.kirby.unsw.edu.au